CLINICAL TRIAL: NCT01686126
Title: A Phase II Randomised Clinical Trial of Mirena® ± Metformin ± Weight Loss Intervention in Patients With Early Stage Cancer of the Endometrium
Brief Title: Improving the Treatment for Women With Early Stage Cancer of the Uterus
Acronym: feMMe
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Queensland Centre for Gynaecological Cancer (Other Government)
Collaborators: The University of Queensland (Other); Queensland University of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: feMMe
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Complex Endometrial Hyperplasia With Atypia; Grade 1 Endometrial Endometrioid Adenocarcinoma
Keywords: endometrial hyperplasia; endometrial adenocarcinoma; Gynecological Cancer
MeSH Terms: conditions — Endometrial Hyperplasia | interventions — Levonorgestrel; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mirena + Metformin (Experimental): Metformin tablets, 500mg twice daily orally, 6 months Levonorgestrel (Mirena®) 52mg Intrauterine drug delivery system, 6 months
  Interventions: Drug: Levonorgestrel; Drug: Metformin
- Mirena (Experimental): Levonorgestrel (Mirena®) 52mg Intrauterine drug delivery system, 6 months
  Interventions: Drug: Levonorgestrel
- Mirena + Weight Loss Intervention (Experimental): Levonorgestrel (Mirena®) 52mg Intrauterine drug delivery system, 6 months Weight Loss Intervention will be delivered via Weight Watchers
  Interventions: Drug: Levonorgestrel

INTERVENTIONS:
Drug: Levonorgestrel — Intrauterine device
  Other Names: Mirena
Drug: Metformin — oral medication
  Arms: Mirena + Metformin

SUMMARY:
Currently the standard treatment for early stage endometrial cancer or endometrial hyperplasia with atypia is a total hysterectomy (an operation to remove the uterus) and removal of both ovaries. While highly effective, this surgery carries significant side effects for:

* young women who still wish to have children and would lose fertility; and
* women with one or more disorders (or diseases) in addition to the early stage endometrial cancer or endometrial hyperplasia with atypia and/or morbid obesity who are at risk for surgical complications making surgery unsafe.

This study will access a new approach to the treatment of endometrial cancer to spare women of having to undergo major surgery that may be unwanted or unnecessary.

Mirena is approved in Australia for contraception, to treat heavy bleeding, and to prevent thickening of the lining of the uterus (endometrial hyperplasia) during oestrogen replacement therapy (HRT). However it is not approved to treat early stage endometrial cancer or endometrial hyperplasia with atypia. This research project will test to see if Mirena is an effective treatment for early stage endometrial cancer and endometrial hyperplasia with atypia.

Metformin is approved in Australia to treat Diabetes. However it is not approved to treat early stage endometrial cancer or endometrial hyperplasia with atypia. Therefore, it is an experimental treatment for early stage endometrial cancer and endometrial hyperplasia with atypia. This means that it must be tested to see if it is an effective treatment for early stage endometrial cancer and endometrial hyperplasia with atypia.

Weight loss interventions are feasible and safe, and already being implemented by gynaecologic oncologist to make women eligible for surgery. Weight loss of 7% body weight induces a large biological effect (for example reduces incidence of diabetes by 58%, and hypertension by 26%).

ELIGIBILITY:
Inclusion Criteria:

1. Females with a BMI > 30 kg/m2 wishing to retain fertility or females who are at high risk of surgical complications due to co-morbidities or obesity
2. Over 18 years of age at time of randomisation
3. Histologically confirmed complex endometrial hyperplasia with atypia or grade 1 endometrioid endometrial adenocarcinoma on a curette or endometrial biopsy
4. CT or MRI scan of pelvis, abdomen and chest (or chest X-Ray) suggesting the absence of extrauterine disease
5. Myometrial invasion on MRI of not more than 50%, for women with histologically confirmed Endometrial Cancer only (for women who are unable to fit into an MRI machine inclusion into trial is at investigators discretion)
6. No lymph vascular invasion on curetting or pipelle, if able to be assessed on sample
7. Serum CA125 ≤ 30 U/mL
8. No hypersensitivity or contraindications for Mirena
9. Ability to comply with endometrial biopsies at specified intervals
10. Negative serum or urine pregnancy test in pre-menopausal women and women < 2 years after the onset of menopause
11. Creatinine < 150µmol/L (1.7 mg/dL) to be randomised into Mirena + Metformin arm (can still be eligible to be randomised to Mirena only or Mirena + Weight Loss, see section 5.4 Other Eligibility Criteria Considerations)

Exclusion Criteria:

1. ECOG performance status > 3
2. Grade 1 endometrioid adenocarcinoma of the endometrium with myometrial invasion deeper than 50% on MRI or any patients with grade 2 or grade 3 endometrioid adenocarcinoma
3. Histological (cell) type other than endometrioid adenocarcinoma (sarcomas or high risk endometrial e.g. papillary serous, clear cell)
4. Pregnant or planning to become pregnant during trial period
5. Has had prior treatment or undergoing current treatment for EAC or EHA
6. Patients with a history of pelvic or abdominal radiotherapy
7. Unwilling to have additional endometrial biopsies or curettes and unable to attend three monthly clinical assessments
8. Unable to provide informed consent
9. Unable or unwilling to complete questionnaires
10. Evidence of extrauterine spread on medical imaging
11. Congenital or acquired uterine anomaly which distorts the uterine cavity
12. Acute pelvic inflammatory disease
13. Conditions associated with increased susceptibility to infections with microorganisms (e.g., AIDS, leukaemia, IV drug abuse) according to the patients Medical History
14. Genital actinomycosis
15. Current other cancer, except low grade malignancies that do not require any systemic treatment or treatment to the pelvis
16. Breastfeeding mothers
17. Mirena inserted greater than 12 weeks before randomisation/enrolment
18. Previous use of Mirena within the last 5 years from randomisation/enrolment
19. Contraindications to both Metformin and weight loss

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 6 months

SECONDARY OUTCOMES:
Predict the response to treatment | 6 months
  To predict the response to treatment through blood and tissue molecular biomarkers and to increase our molecular understanding of the biological pathogenesis of "early" EAC.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Obermair, Study Chair — Queensland Centre for Gynaecological Cancer
Locations (17):
- Australia (13):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - The Wesley Hospital, Auchenflower, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Mater Health Services, Brisbane, South Brisbane, Queensland
  - Mater Private Hospital, South Brisbane, Queensland
  - Gold Coast Hospital, Southport, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Women's Hospital, Carlton, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - King Edward Memorial Hospital for Women, Perth, Western Australia
  - St John of God Hospital, Subiaco, Western Australia
- New Zealand (4):
  - Auckland City Hospital, Auckland
  - Middlemore Hospital, Auckland
  - Christchurch Women's Hospital, Christchurch
  - Wellington Hospital, Wellington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Janda M, Robledo KP, Gebski V, Armes JE, Alizart M, Cummings M, Chen C, Leung Y, Sykes P, McNally O, Oehler MK, Walker G, Garrett A, Tang A, Land R, Nicklin JL, Chetty N, Perrin LC, Hoet G, Sowden K, Eva L, Tristram A, Obermair A. Complete pathological response following levonorgestrel intrauterine device in clinically stage 1 endometrial adenocarcinoma: Results of a randomized clinical trial. Gynecol Oncol. 2021 Apr;161(1):143-151. doi: 10.1016/j.ygyno.2021.01.029. PMID 33762086